CLINICAL TRIAL: NCT00533624
Title: Head to Head Comparison of Myfortic vs. Cellcept in the Treatment of Kidney Transplant Recipients Using Our Current Center Standardized Concomitant Immunosuppressive Protocol
Brief Title: Myfortic vs. Cellcept in Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A-US10
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: End Stage Renal Disease
Keywords: Gastrointestinal toxicity
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Myfortic (Active Comparator): Myfortic Group: Myfortic® 1,440 mg/day in two divided doses (induced with either the IL-2 receptor inhibitors or thymoglobulin). Tacrolimus will be dosed to 12-hour trough levels of 8-10 ng/ml. Methylprednisolone is to be given as per our center protocols, weaning to dose levels of <0.1 mg/kg by 3-6 months post-operatively.
  Interventions: Drug: Mycophenolate Sodium Delayed Release Tablets
- 2. Cellcept (Active Comparator): Cellcept® 2,000 mg/day, in divided doses (induced with either the IL-2 receptor inhibitors or thymoglobulin). Tacrolimus will be dosed to 12-hour trough levels of 8-10 ng/ml. Methylprednisolone is to be given as per our center protocols, weaning to dose levels of <0.1 mg/kg by 3-6 months post-operatively.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Sodium Delayed Release Tablets — Myfortic® 1,440 mg/day
  Arms: 1: Myfortic
Drug: Mycophenolate Mofetil — Cellcept® 2,000 mg/day
  Other Names: Cellcept®
  Arms: 2. Cellcept

SUMMARY:
The comparison the incidence of G.I. toxicity between Myfortic® vs. Cellcept® in 150 sequential patients, in which 75 will be randomized to Cellcept® and 75 to Myfortic® in first and second living or deceased donor renal transplant recipients.

DETAILED DESCRIPTION:
Purpose and Description:

The purpose of the study is to determine if gastrointestinal toxicity of an anti-rejection medication Myfortic® (mycophenolic acid delayed release) is less than equivalent doses of a similar anti-rejection medication Cellcept® (mycophenolate mofetil, MMF) in patients receiving their first or second kidney transplant from cadaver or living donors.

This study consist of two randomized groups, 75 patients given 3 doses of Thymoglobullin (Group I) vs. 75 patients given 3 doses of Thymoglobulin and 2 doses of Basiliximab (Group II).

Our standard maintenance protocol dosing of tacrolimus, IMPDH inhibitor (vide infra) and one week course of corticosteroids.

Patients will be randomized to receive Myfortic® 1,440 mg/day vs. Cellcept® 2,000 mg/day, each in two divided doses (induced with either the IL-2 receptor inhibitors or thymoglobulin). Tacrolimus will be dosed to 12-hour trough levels of 8-10 ng/ml. Methylprednisolone is to be given as per our center protocols, weaning to dose levels of <0.1 mg/kg by 3-6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been fully informed and has signed a dated IRB approval informed consent form and is willing to follow study procedures for the extent of the study (12 months). Parent or legal guardian must provide written consent for patients <18 years of age.
2. Age 18-75 years.
3. Weight > 40 kg.
4. Primary or secondary renal allograft: living or deceased donor.
5. Negative standard crossmatch for T cells.
6. Women of childbearing potential will be required to have a negative qualitative serum pregnancy test and agree to use an adequate method of contraception for the study duration.
7. Males and females are to be studied equivalently as they become available for transplantation using these criteria.

Exclusion Criteria:

1. Patient has previously received or is receiving an organ transplant other than a kidney.
2. Patient is receiving an ABO incompatible donor kidney.
3. Recipient or donor is seropositive for human immunodeficiency (HIV), Hepatitis C viruses, or Hepatitis B virus antigenemia.
4. Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully, or carcinoma in situ of the cervix that has been treated successfully.
5. Patients with significant liver disease, defined as having during the past 28 days continuously elevated AST (SGOT) and/or ALT (SGPT) levels greater than 3 times the upper value of the normal range of this center.
6. Patient has uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or an active peptic ulcer or any other unstable medical condition that could interfere with study objectives.
7. Patient is currently participating in another clinical trial of an investigational drug in the 30 days prior to transplant.
8. Patient will be receiving any immunosuppressive agent other than those prescribed in the study.
9. Patient is unable to take medications orally or via nasogastric tube by the morning of the second day following completion of the transplant procedure (i.e., skin closure) (Group I only).
10. Patient is receiving or may require warfarin, fluvastatin, or herbal supplements during the study.
11. Concurrent use of astemizole, pimozide, cisapride, terfenadine, or ketoconazole.
12. Patient has a known hypersensitivity to tacrolimus, thymoglobulin, IL-2 receptor inhibitor monoclonal antibodies, sirolimus, MMF, Myfortic®, or corticosteroids.
13. Patient is pregnant or lactating.
14. Patients with a screening/baseline (or within 96 hours of transplant) total white blood cell count <4000/mm3; platelet count <100,000/mm3; fasting triglycerides >400 mg/dl (>4.6 mmol/L); fasting total cholesterol >300 mg/dl (>7.8 mmol/L); fasting HDL-cholesterol <30 mg/dl; fasting LDL-cholesterol >200 mg/dl.
15. Patient is unlikely to comply with the visits scheduled in the protocol.
16. Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.

If tacrolimus cannot be instituted for longer than 5 days postoperatively.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Observation of G.I. toxicity (nausea, vomiting, or diarrhea). One year patient and graft survival after initiation of study agent.Incidence of biopsy-proven acute rejection (vide infra). 4. Incidence of chronic allograft nephropathy (vide infra). | 1 year

SECONDARY OUTCOMES:
Incidence of AE: Infections, malignancies (including PTLD), thromboembolic events, hyperlipidemia and leuko and thrombocytopenia, cytokine release syndrome with induction antibody agents, wound healing and lymphocele, post-tx diabetes. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George W Burke, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

REFERENCES:
- [Derived] Ciancio G, Gaynor JJ, Sageshima J, Roth D, Kupin W, Guerra G, Tueros L, Zarak A, Hanson L, Ganz S, Chen L, Ruiz P, Livingstone AS, Burke GW 3rd. Machine perfusion following static cold storage preservation in kidney transplantation: donor-matched pair analysis of the prognostic impact of longer pump time. Transpl Int. 2012 Jan;25(1):34-40. doi: 10.1111/j.1432-2277.2011.01364.x. Epub 2011 Oct 8. PMID 21981661